CLINICAL TRIAL: NCT01463891
Title: Post-marketing Surveillance for the Clinical Safety and Effectiveness of Eribulin Mesylate in Patients With Inoperable or Recurrent Breast Cancer
Brief Title: Post-marketing Surveillance for the Clinical Safety and Effectiveness of Eribulin Mesylate in Patients With Inoperable or Recurrent Breast Cancer (Study HAL01S)
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: HAL01S
Record Dates: First submitted 2011-09-29; First posted 2011-11-02 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2016-12

CONDITIONS: Inoperable or Recurrent Breast Cancer
Keywords: Eribulin Mesylate; inoperable or recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Eribulin Mesylate
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate — The usual adult dose of eribulin mesylate is 1.4 mg/m^2 (body surface area) administered intravenously over 2 to 5 minutes, once daily once a week. Treatment shall be continued for 2 consecutive weeks followed by a third week of drug cessation. With each cycle lasting 3 weeks, the treatment shall be repeated. The dose may be reduced, depending on the condition of the individual patient.

SUMMARY:
To investigate of the clinical safety and effectiveness of eribulin mesylate in patients with inoperable or recurrent breast cancer

ELIGIBILITY:
Inclusion criteria :

* Inoperable breast cancer
* Recurrent breast cancer

Exclusion criteria :

* Corresponding to contraindication of eribulin mesylate
* Not applicable to indications of eribulin mesylate
* Not applicable to aggravation or recurrence of breast cancer in patients who have previously been treated with anthracycline and/or taxane antitumor drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals and clinics in Japan
Sampling Method: Non-Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2011-07-19 (Actual); Primary Completion 2012-12-26 (Actual); Study Completion 2013-11-27 (Actual)

PRIMARY OUTCOMES:
Effectiveness Diagnosed by Imaging | 1 year
  Effectiveness diagnosed by imaging, is based on Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. Defined as:
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to less than10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
  * Not Evaluable (NE).

CONTACTS AND LOCATIONS:
Overall Officials: Toshiyuki Matsuoka, Study Director — Drug Fostering and Evolution Cordination Department, Eisai Co., Ltd.
Locations (223):
- Japan (223):
  - Anjo, Aichi-ken
  - Inazawa, Aichi-ken
  - Kariya, Aichi-ken
  - Komaki, Aichi-ken
  - Nagakute, Aichi-ken
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Seto, Aichi-ken
  - Tahara, Aichi-ken
  - Toyohashi, Aichi-ken
  - Daisen, Akita
  - Yokote, Akita
  - Goshogawara, Aomori
  - Hirosaki, Aomori
  - Kuroishi, Aomori
  - Misawa, Aomori
  - Mutsu, Aomori
  - Asahi, Chiba
  - Funabashi, Chiba
  - Ichihara, Chiba
  - Ichikawa, Chiba
  - Kashiwa, Chiba
  - Kimitsu, Chiba
  - Matsudo, Chiba
  - Sakura, Chiba
  - Matsuyama, Ehime
  - Niihama, Ehime
  - Iizuka, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Omuta, Fukuoka
  - Yame, Fukuoka
  - Yanagawa, Fukuoka
  - Minamisoma, Fukushima
  - Nihommatsu, Fukushima
  - Ena, Gifu
  - Hashima, Gifu
  - Minokamo, Gifu
  - Ōgaki, Gifu
  - Sekimachi, Gifu
  - Tajimi, Gifu
  - Takayama, Gifu
  - Maebashi, Gunma
  - Ōta, Gunma
  - Shibukawa, Gunma
  - Takasaki, Gunma
  - Aki, Hiroshima
  - Fukuyama, Hiroshima
  - Hatsukaichi, Hiroshima
  - Higashihiroshima, Hiroshima
  - Kure, Hiroshima
  - Mihara, Hiroshima
  - Onomichi, Hiroshima
  - Abashiri, Hokkaido
  - Asahikawa, Hokkaido
  - Date, Hokkaido
  - Eniwa, Hokkaido
  - Hakodate, Hokkaido
  - Kitahiroshima, Hokkaido
  - Kitami, Hokkaido
  - Kushiro, Hokkaido
  - Muroran, Hokkaido
  - Obihiro, Hokkaido
  - Sapporo, Hokkaido
  - Shibetsu, Hokkaido
  - Akashi, Hyōgo
  - Amagasaki, Hyōgo
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Toyooka, Hyōgo
  - Higashiibaraki, Ibaraki
  - Inashiki, Ibaraki
  - Kamisu, Ibaraki
  - Kasama, Ibaraki
  - Koga, Ibaraki
  - Moriya, Ibaraki
  - Tsukuba, Ibaraki
  - Ushiku, Ibaraki
  - Kahoku, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Komatsu, Ishikawa-ken
  - Nomi, Ishikawa-ken
  - Takamatsu, Kagawa-ken
  - Akune, Kagoshima-ken
  - Chigasaki, Kanagawa
  - Ebina, Kanagawa
  - Isehara, Kanagawa
  - Kamakura, Kanagawa
  - Kawasaki, Kanagawa
  - Odawara, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Arao, Kumamoto
  - Tamana, Kumamoto
  - Kōtari, Kyoto
  - Ise, Mie-ken
  - Matsusaka, Mie-ken
  - Suzuka, Mie-ken
  - Tsu, Mie-ken
  - Yokkaichi, Mie-ken
  - Murata, Miyagi
  - Ōsaki, Miyagi
  - Sendai, Miyagi
  - Iida, Nagano
  - Komagane, Nagano
  - Matsumoto, Nagano
  - Saku, Nagano
  - Suwa, Nagano
  - Shimabara, Nagasaki
  - Ikoma, Nara
  - Kashihara, Nara
  - Yamatotakada, Nara
  - Minamiuonuma, Niigata
  - Kurashiki, Okayama-ken
  - Maniwa, Okayama-ken
  - Tamano, Okayama-ken
  - Wake, Okayama-ken
  - Naha, Okinawa
  - Nakagami, Okinawa
  - Shimajiri, Okinawa
  - Tomigusuku, Okinawa
  - Urasoe, Okinawa
  - Higashiosaka, Osaka
  - Hirakata, Osaka
  - Ibaraki, Osaka
  - Izumiōtsu, Osaka
  - Katano, Osaka
  - Neyagawa, Osaka
  - Sayama, Osaka
  - Takatsuki, Osaka
  - Yao, Osaka
  - Karatsu, Saga-ken
  - Fujimino, Saitama
  - Fukaya, Saitama
  - Hidaka, Saitama
  - Hiki, Saitama
  - Kawaguchi, Saitama
  - Kumagaya, Saitama
  - Toda, Saitama
  - Tokorozawa, Saitama
  - Kusatsu, Shiga
  - Ōtsu, Shiga
  - Rittō, Shiga
  - Izumo, Shimane
  - Matsue, Shimane
  - Fujieda, Shizuoka
  - Fujinomiya, Shizuoka
  - Gotemba, Shizuoka
  - Hamamatsu, Shizuoka
  - Izunokuni, Shizuoka
  - Numazu, Shizuoka
  - Shimada, Shizuoka
  - Sunto, Shizuoka
  - Ashikaga, Tochigi
  - Oyama, Tochigi
  - Adachi City, Tokyo
  - Akishima, Tokyo
  - Bunkyo, Tokyo
  - Chiyoda City, Tokyo
  - Chūō, Tokyo
  - Fuchū, Tokyo
  - Fussa, Tokyo
  - Hachiōji, Tokyo
  - Hino, Tokyo
  - Katsushika-ku, Tokyo
  - Kita-ku, Tokyo
  - Koto, Tokyo
  - Machida, Tokyo
  - Meguro City, Tokyo
  - Minato, Tokyo
  - Mitaka, Tokyo
  - Nerima City, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya City, Tokyo
  - Shibuya City, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku, Tokyo
  - tabashi City, Tokyo
  - Tachikawa, Tokyo
  - Taitō City, Tokyo
  - Tama, Tokyo
  - Kurayoshi, Tottori
  - Yonago, Tottori
  - Nakaniikawa, Toyama
  - Namerikawa, Toyama
  - Oyabe, Toyama
  - Takaoka, Toyama
  - Tsuruoka, Yamagata
  - Hagi, Yamaguchi
  - Iwakuni, Yamaguchi
  - Nagato, Yamaguchi
  - Shimonoseki, Yamaguchi
  - Chūō, Yamanashi
  - Kofu, Yamanashi
  - Minamikoma, Yamanashi
  - Aomori
  - Chiba
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Hiroshima
  - Kagoshima
  - Kochi
  - Kumamoto
  - Kyoto
  - Miyazaki
  - Nagano
  - Nagasaki
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Shizuoka
  - Tokushima
  - Tottori
  - Toyama

REFERENCES:
- [Result] Watanabe J, Ito Y, Ohsumi S, Mizutani M, Tashiro H, Sakurai K, Takahashi M, Saito T, Tsurutani J, Mukai H, Yoshinami T, Takao S, Yamamoto Y, Matsuoka T, Iwase H, Iwata H, Nakamura S, Saeki T. Safety and effectiveness of eribulin in Japanese patients with locally advanced or metastatic breast cancer: a post-marketing observational study. Invest New Drugs. 2017 Dec;35(6):791-799. doi: 10.1007/s10637-017-0486-4. Epub 2017 Jun 29. PMID 28660549